CLINICAL TRIAL: NCT03289078
Title: Evaluation of Functional Improvement After Spa Therapy in Fontcaude Center, for Knee Osteoarthritis
Brief Title: Evaluation of Functional Improvement After Spa Therapy in Fontcaude Center
Acronym: FONTCAUDE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No financing
Sponsor: University Hospital, Montpellier (Other)
Collaborators: FONTCAUDE's Vichy SPA center, Juvignac (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 9846
Record Dates: First submitted 2017-09-18; First posted 2017-09-20 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thermal care (Experimental): Spa Treatment realised daily 6 days a week during 18 days
  Interventions: Other: Spa Treatment
- Standard Care (No Intervention): Usual care

INTERVENTIONS:
Other: Spa Treatment — The spa treatments will be realised daily 6 days a week and during 18 days. The care will be provided is : Swimming pool of mobilization by physical therapist (20 minutes daily, Cataplasms (10 minutes daily), Shower in the jet (10 minutes daily), Shower under affusion (10 minutes daily)
  Arms: Thermal care

SUMMARY:
Evaluation of functional improvement after spa therapy in Fontcaude center, for knee osteoarthritis Background. Knee osteoarthritis is the first indication of spa therapy in rheumatology. This therapeutic represents a non pharmacological treatment and is recommended by OARSI.

In order to obtain agreement for spa therapy, the center Fontcaude, needs to show clinical improvement for patients, as demonstrated in the Thermarthrose study. This center is near Montpellier and could improve patients localised in this area.

DETAILED DESCRIPTION:
Methods: randomised prospective clinical trial of patients with knee osteoarthritis.

The spa therapy group received 18 days of therapy over 3 weeks. Patients in the control group received 18 days of therapy over 3 weeks after the 6-month follow-up visit.

Follow-up was at 3 and 6 months, by a visit to the examination.

The hypothesis of our study is to demonstrate clinical improvement at six months. The main endpoint is the number of patients achieving minimal clinically important improvement (MCII) at 6 months, defi ned as ≥19.9 mm on the visual analogue pain scale and/or ≥9.1 points in a normalised Western Ontario and McMaster Universities osteoarthritis index function score.

ELIGIBILITY:
Inclusion criteria:

* Patient aged 40 to 75 years with radiologic and gonarthrosis radiologic et painful gonarthrosis, unilateral ou bilateral, whatever is the radiographic stage
* Patient presenting a EVA ≥3 with a corresponding radiology at least of 1year
* Patient affiliated with a social security system

Exclusion criteria:

* Realization of a water cure in the last 6 months
* Infiltration of the knee of less than 3 months
* Impossibility to sign the informed consent or which for reasons geographical, social or psychological could not be regularly followed,
* Person major placed under guardianship or trusteeship,
* Private person of freedom by court or administrative order, nobody being the object of a legal protective measure,
* Patient already included in an interventional clinical protocol,
* Pregnant women
* Contraindication in the water cure:

  * Severe change of the general state or debilitating afflictions
  * Acute affections and pushed acute(sharp) of the chronic affections
  * Grave cardiac insufficiency, unstable arterial high blood pressure
  * Severe renal or hepatic insufficiency
  * Not healed cutaneous hurts
  * Contagious or evolutionary diseases
  * Evolutionary Cancers
  * Current immunomodulator or immunosupressor Treatment, waves of inflammation.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Achievement of minimal clinically important improvement (MCII) at 6 months | 30 months
  The main endpoint is the number of patients achieving minimal clinically important improvement (MCII) at 6 months, defined as ≥19.9 mm on the visual analogue pain scale and/or ≥9.1 points in a normalised Western Ontario and McMaster Universities osteoart

SECONDARY OUTCOMES:
Achievement of minimal clinically important improvement (MCII) at 3 months | 30 months
  The second outcome measure is the number of patients achieving minimal clinically important improvement (MCII) at 3 months, defi ned as ≥19.9 mm on the visual analogue pain scale and/or ≥9.1 points in a normalised Western Ontario and McMaster Universities osteoarthritis index function score, and also the safety.

CONTACTS AND LOCATIONS:
Overall Officials: Isabel TAVARES, PH, Principal Investigator — CHU de Montpellier

IPD SHARING:
Plan to Share IPD: No